CLINICAL TRIAL: NCT05758948
Title: Detection of Germline and Somatic Pathogenic Variants in Patients With de Novo Metastatic Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: Hellenic Society of Medical Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: TRANS_DNM_17
Record Dates: First submitted 2023-02-15; First posted 2023-03-08 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood and Formalin-Fixed Paraffin-Embedded (FFPE) tissue specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with de novo metastatic breast cancer: Blood and tissue sample from patients diagnosed with DN-MBC will be analyzed using next generation sequencing (NGS)
  Interventions: Diagnostic Test: NGS in blood and Formalin-Fixed Paraffin-Embedded (FFPE) tissue

INTERVENTIONS:
Diagnostic Test: NGS in blood and Formalin-Fixed Paraffin-Embedded (FFPE) tissue — In patients with denovo metastatic breast cancer blood and tissue sample will be collected and then further analysed using NGS in order to detect somatic and germline pathogenic variants

SUMMARY:
To determine somatic and germline pathogenic variants in patients with denovo metastatic breast cancer in order to map the molecular/genetic characteristics of DN- MBC aiming in comprehending the biology and highlighting potential novel treatment options for the disease.

DETAILED DESCRIPTION:
The value of this study is based on the fact that DN-MBC is rare, seems to be different from early and relapsed breast cancer and has not been studied as distinct disease. To achieve the objective of this study blood and tissue sample from patients diagnosed with DN-MBC will be further analyzed using next generation sequencing (NGS), in order to map the molecular/genetic characteristics of DN-MBC and to detect germline and somatic pathogenic variants. All the results will be associated with the clinicopathological characteristics of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent for the provision of the biological material for research purposes
2. Diagnosis of de novo MBC (histologically confirmed)
3. Age >18 years
4. Blood samples
5. Tumor tissue block from at least on disease site, primary (preferably) or metastatic

Exclusion Criteria:

Inadequate MBC tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients will be selected from community or academic or private hospitals
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 1998-07-05 (Actual); Primary Completion 2010-10-05 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with somatic pathogenic variants in denovo metastatic breast cancer | up to 12 months
Number of participants with germline pathogenic variants in denovo metastatic breast cancer | up to 12 months

SECONDARY OUTCOMES:
Definition of the somatic pathogenic variants measured with Next Generation Sequencing | up to 12 months
Collection of clinicopathological characteristics of the included patients from patient's medical file | up to 12 months
Definition of the germline pathogenic variants measured with Next Generation Sequencing | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: EVANGELIA MOIROGIORGOU, Principal Investigator — YGEIA Hospital
Locations (1):
- Evangelia Moirogiorgou, Athens, Greece